CLINICAL TRIAL: NCT07076524
Title: The Relationship Between Oral and Suprahyoid Muscle Wasting and Dysphagia in Critically Ill Patients
Brief Title: MuScle WastIng and DysphaGia iN CriticAlly IlL Patients (SIGNAL)
Acronym: SIGNAL
Status: Recruiting | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 348596; G-002784 (Other Grant/Funding Number: Barts Charity)
Record Dates: First submitted 2025-05-22; First posted 2025-07-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Dysphagia; Muscle Wasting in Critically Ill; Swallowing Disorders
Keywords: dysphagia; critical illness; swallowing disorders; muscle wasting
MeSH Terms: conditions — Critical Illness; Deglutition Disorders; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to find out how muscle wasting in the mouth and throat affects swallowing (dysphagia) in adults who are critically ill and being treated in intensive care units.

The main aims of this research study are to understand: how much and how quickly the oral and suprahyoid muscles waste in critically ill participants, and whether muscle wasting causes problems with swallowing. The investigators will compare critically ill participants with non-critically ill participants to determine if muscle wasting is linked to swallowing problems.

In this study, participants will have the size and strength of their mouth and throat muscles measured at four different times during their critical care admission and hospital stay. Tests will also be performed to check how well and how safely participants can swallow. Tongue strength will be measured, and participants will answer questions about their experience with swallowing and eating using patient-reported outcome measures.

This study may help identify better ways to diagnose and treat swallowing problems in people who are critically ill, to support safe eating and drinking and promote faster recovery.

DETAILED DESCRIPTION:
Background:

Dysphagia is a common and serious complication among critically ill patients admitted to intensive care units (ICUs). Up to 62% of patients who require mechanical ventilation experience dysphagia, which can lead to aspiration pneumonia, malnutrition, longer hospital stays, and increased mortality. Muscle wasting is a known consequence of critical illness and is associated with poor functional outcomes. The contribution of oral and suprahyoid muscle wasting to dysphagia in critically ill participants is poorly understood. This study aims to prospectively evaluate muscle wasting and its impact on swallowing function in critically ill adults.

Ethical Approval:

This study has Research Ethics Committee and Health Research Authority approval.

Study Objectives:

Primary Objective:

To measure the extent and rate of change in the cross-sectional area of the oral and suprahyoid muscles in critically ill adults using bedside ultrasound at four time points, and to relate these changes to swallowing physiology and safety.

Secondary Objectives:

To compare muscle mass and swallowing function between critically ill and non-critically ill participants.

To measure electrophysiological features of swallowing muscles using high-definition surface electromyography.

To assess patient-reported outcomes related to swallowing and eating.

To compare changes in the rectus femoris (thigh) muscle to those in the oral and suprahyoid muscles as a reference for general muscle wasting.

Study Design:

This is a prospective observational study. Critically ill participants admitted to the ICU will be recruited and compared with non-critically ill controls. The study includes repeated measures of muscle size and swallowing function over time.

Study Procedures:

Ultrasound Assessments:

The cross-sectional area of the tongue, geniohyoid, mylohyoid, and anterior belly of digastric muscles will be measured using bedside ultrasound at four time points during the participant's ICU stay. The rectus femoris muscle will also be measured as a reference for general muscle wasting.

Swallowing Evaluation:

Instrumental assessments of swallowing physiology and safety will be performed using gold standard assessments (e.g., videofluoroscopy or fiberoptic endoscopic evaluation of swallowing).

Tongue Strength:

Tongue strength will be measured using tongue dynamometry.

Electromyography:

High-definition surface electromyography will assess muscle activation patterns at rest and during swallowing.

Patient-Reported Outcomes:

Participants will complete patient reported outcome measures on swallowing, eating, and quality of life.

Data Management and Quality Assurance:

Data will be collected and managed according to Good Clinical Practice (GCP) and UK data protection regulations. Data will be collected using an online database (RedCap). Monitoring and auditing will be conducted by the sponsor to ensure protocol adherence and data integrity.

Sample Size and Statistical Analysis:

The sample size is calculated to detect clinically meaningful differences in muscle wasting and swallowing outcomes, based on expected rates in critically ill patients. Sample size was calculated based on a proof-of-conduct study completed by the investigators.

The primary analysis will use mixed-effects models to evaluate changes in muscle size and their association with swallowing function over time. Secondary analyses will compare critically ill patients with non-critically ill controls and explore associations between muscle wasting, swallowing outcomes, and patient-reported measures. Missing data will be addressed using appropriate statistical methods, such as multiple imputation or sensitivity analyses, as detailed in the statistical analysis plan.

Safety and Adverse Event Reporting:

The study involves only non-invasive assessments; risks are minimal and mainly relate to patient discomfort during swallowing tests. Adverse events and serious adverse events will be monitored and reported according to regulatory requirements.

Patient and Public Involvement:

Patients with experience of dysphagia in critical care contributed to the design of the study and the selection of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Receiving mechanical ventilation via endotracheal tube and/or tracheostomy. Expected to receive ventilation for at least 72 hours.
* Expected to survive admission and spend more than 7 days in the intensive care unit.

Control participants

* Adults >18 years
* Receiving ward-based care.
* Expected to survive hospital admission. Present with a primary medical diagnosis of acute medical or surgical illness, not requiring critical care admission.

Exclusion Criteria:

Applies to both critically ill and control participants.

* Pregnancy
* Patients with a diagnosis of a primary neuromuscular pathology (e.g., motor neurone disease), central nervous system disease (e.g., stroke, Guillain barre), traumatic brain injury, connective tissue disease (e.g., scleroderma), head and neck cancer, previous surgery or radiotherapy to the head and neck.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients and non-critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Measure the extent and rate of muscle wasting | Day 1, 3, 7 and 10 of intensive care unit admission
  To measure the extent and rate of change in cross-sectional area of the oral and suprahyoid muscles in critically ill adults using bedside ultrasound across four time points. The extent and rate of muscle wasting will be assessed by measuring the change in cross-sectional area (mm²) of the oral and suprahyoid muscles using bedside ultrasound.
Relate muscle wasting to swallow physiology and safety | Following day 10 ultrasound or when the patient is extubated and clinically appropriate for swallow assessment
  To correlate changes in cross-sectional area to swallow physiology and safety in critically ill patients, using instrumental swallowing evaluations and tongue strength. To quantify the change in size of the oral and suprahyoid muscles, the cross-sectional area (mm²) will be measured using bedside ultrasound. Swallowing physiology and safety will be assessed using instrumental swallowing evaluations (e.g., Fiberoptic Endoscopic Evaluation of Swallowing (FEES)).The correlation coefficient (e.g., Pearson's or Spearman's r) between ultrasound-measured muscle cross-sectional area and instrumental swallowing assessment scores (e.g., the Penetration Aspiration Scale) will be used.

SECONDARY OUTCOMES:
Measure electrophysiological features of swallow muscle activity | Day 1, 3, 7 and 10 of intensive care unit admission
  To measure the electrophysiological features of swallowing muscles using high definition surface electromyography in critically ill and non-critically ill patients. Electrophysiological features of swallowing-related muscles will be measured. Parameters will include average root mean square amplitude, symmetry of muscle activation, and duration of muscle activity during swallowing tasks.
Compare relationship between muscle mass and swallow physiology | Day 1, 3, 7 and 10 ultrasound assessments, swallow evaluation completed following day 10 ultrasound or when patient is extubated and clinically appropriate
  To compare the relationship between muscle mass and swallow physiology in critically ill patients and non-critically ill patients. The correlation between muscle mass and swallow physiology will be assessed. Muscle mass will be measured using ultrasound cross-sectional area (cm²) of the oral and suprahyoid muscles at four time points: Day 1, Day 3, Day 7, and Day 10 of ICU admission. Swallow physiology will be evaluated using instrumental evaluation (e.g., flexible endoscopic evaluation of swallow) and the following scales: Penetration-Aspiration Scale, Yale Pharyngeal Residue Severity Rating Scale and the Dynamic Imaging Grade of Swallow Toxicity) whichever occurs first, and when the patient is deemed clinically appropriate for assessment. The primary outcome will be the correlation coefficient (e.g., Pearson's or Spearman's r) between ultrasound-measured muscle mass (cm²) and swallow physiology scores.
Patient reported outcomes: Sydney Swallow Questionnaire | Within two weeks of day 10 ultrasound measurement or when clinically appropriate (e.g., ICU delirium resolved if present), up to 1 month
  Patient-reported severity of dysphagia symptoms will be assessed using the Sydney Swallow Questionnaire (SSQ), with the total score ranging from 0 to 1700, where higher scores indicate greater symptom severity.
Patient reported outcomes: Swallowing Quality of Life (SWAL-QoL) Score | Within two weeks of day 10 ultrasound measurement or when clinically appropriate (e.g., ICU delirium resolved if present), up to 1 month
  Patient-reported swallowing-related quality of life will be assessed using the Swallowing Quality of Life (SWAL-QoL) questionnaire, a 44-item instrument producing a total score from 0 to 100, where higher scores reflect better quality of life.
Patient reported outcomes: Functional Oral Intake Scale | Within two weeks of day 10 ultrasound measurement or when clinically appropriate (e.g., ICU delirium resolved if present), up to 1 month
  Functional oral intake level will be measured using the Functional Oral Intake Scale (FOIS), a 7-point ordinal scale ranging from 1 (nothing by mouth) to 7 (total oral diet with no restrictions), where higher scores represent greater functional intake.
Patient reported outcomes: Eating Assessment Tool-10 (EAT-10) | Within two weeks of day 10 ultrasound measurement or when clinically appropriate (e.g., ICU delirium resolved if present), up to 1 month
  Patient-reported dysphagia symptom burden will be screened using the Eating Assessment Tool-10 (EAT-10), a 10-item instrument with total scores ranging from 0 to 40, where scores of 3 or higher suggest abnormal swallowing.
Compare the extent of muscle wasting in critically ill versus non-critically ill patient | Day 1, 3, 7 and 10 ultrasound evaluation vs single timepoint in non-critically ill patients
  To measure and compare the extent and rate of change in cross-sectional area of the rectus-femoris muscle and the oral and supra-hyoid muscles using bedside ultrasound across four time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided